CLINICAL TRIAL: NCT06759792
Title: Effect of Physical Activity on Eye Hand Coordination in Patient With Strabismus Amblyopia Post Surgery
Brief Title: Physical Activity on Eye Hand Coordination Post Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amany Refaat Mohamed Abdel Wahid (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Amany Refaat Mohamed Abdel Wahid, lecturer at surgery department, faculty of physical therapy, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005409
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Coordination Impairment
Keywords: amblyopia; strabismus; physical therapy; exercises; eye hand coordination
MeSH Terms: conditions — Ataxia; Amblyopia; Strabismus; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eye hand coordination exercise (Experimental): this group will receive therapeutic exercises to improve eye hand coordination post strabismus surgery
  Interventions: Other: eye hand coordination exercises
- traditional eye observation (No Intervention): this group will receive traditional eye observation post strabismus surgery

INTERVENTIONS:
Other: eye hand coordination exercises — exercises to improve eye hand coordination post strabismus surgery
  Arms: eye hand coordination exercise

SUMMARY:
The aim of this study is to determine the effect of physical activity on eye hand coordination in patient with amblyopia after strabismus surgery.

DETAILED DESCRIPTION:
Eye hand coordination is essential to many of everyday activities. Strabismus not only affect vision but also affect eye hand activities and coordination. Through this study the patients will apply physical therapy sessions to improve eye hand coordination for strabismus amblyopic patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients are both males and females.
* Their age will range from (10-14) years.
* Patients received strabismus operation.
* Patients are suffering from strabismic amblyopia
* Patients are suffering from eye hand coordination problems
* Patients will begin the training program after 2 months of operation.
* All types of strabismus surgery will be included.

Exclusion Criteria:

* Patient who didn't complete the physiotherapy training program for 3 months.
* Muscular disorders that will impair performance during training.
* Any organic lesion in the eye.
* Neurological disorders.
* Malignant conditions.
* Psychiatric illness, severe behavior or cognitive disorders.
* Children who can't understand the therapist's instructions and orders
* Amblyopia which is not related to strabismus condition .

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Eye Hand Coordination Test | From enrollment to the end of treatment at 12 weeks
  * Participants throw a ball against the wall with one hand during axillary movements and try to catch it with the other hand.
  * Purpose: To measure hand-eye coordination
  * Equipment required Tennis or baseball, smooth and solid wall, marking belt, stopwtch (optional)
  * Procedure: Place a mark at a certain distance from the wall (2 meters). The person is standing behind the line, facing the wall. The ball will be thrown towards the wall in an underarm motion from one hand and try to catch it with the other hand. Then throw the ball back to the wall and catch it with the original hand. The test can continue for a specified number of attempts or a set
  * period will be 30 seconds.
  * Scoring: This table lists the general scores of the wall throw test based on the number of successful catches in 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Amany R M Abdel Wahid, Doctoral degree, Principal Investigator — lecturer at faculty of physical therapy, Cairo University
Locations (1):
- Cairo University, Giza, Giza Governorate, Egypt